CLINICAL TRIAL: NCT02418780
Title: Tai Chi for Enhancing Motor and Cognitive Function in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: Spaulding Rehabilitation Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Peter Wayne, Assistant Professor of Medicine, Harvard University Faculty of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013P002343
Record Dates: First submitted 2015-04-06; First posted 2015-04-16 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Tai Ji

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi (Experimental): 6-month Tai Chi training program combined with usual medical care
  Interventions: Other: Tai Chi
- Usual Care (No Intervention): Waitlist control group receiving usual medical care alone

INTERVENTIONS:
Other: Tai Chi — 6-month Tai Chi exercise program meeting 2 times per week plus DVD for home practice
  Arms: Tai Chi

SUMMARY:
The purpose of this feasibility study is to preliminarily evaluate the effects of Tai Chi - a mind-body exercise - on motor and cognitive function as well as quality of life in individuals recently diagnosed with Parkinson's disease (PD).

DETAILED DESCRIPTION:
Specific Aim 1: To assess the feasibility of recruiting and retaining individuals with PD into a 6-month randomized controlled trial of Tai Chi exercise.

Specific Aim 2: To collect preliminary data on the efficacy of Tai Chi on improving gait and balance dynamics, physical and cognitive function, exercise activity, self-efficacy, mood, and quality of life in individuals with PD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals recently diagnosed with idiopathic PD (≤ 10 years)
* Limited disease progression
* If taking PD-related medication, willingness to undergo baseline and follow-up testing while off medication
* Willingness to commit to the study protocols and complete Tai Chi program
* Willingness to be videotaped and audio-recorded during testing

Exclusion Criteria:

* Diagnosis of any form of atypical parkinsonism
* History of: stroke, head trauma, brain tumor, brain injury, seizures or other central nervous system condition, orthopedic impairment or other disease that could likely contribute to a gait disturbance or parkinsonism
* Any severe, chronic condition or acute medical event for which participation in exercise programs is contraindicated (e.g. debilitating Rheumatoid Arthritis, history of frequent falls, unhealed fracture)**

  ** Unless the participant is able to obtain formal written approval from his/her treating physician granting permission to participate in our Tai Chi exercise program
* Participation in brain stimulation within the past 3 months
* Family history of seizures or unexplained loss of consciousness
* Current history of dementia or severe psychiatric illness. Patients with mild (non-suicidal) depression and/or anxiety may be included
* Acute illness requiring hospitalization within past 3 months
* History of deep brain stimulation or other brain surgery
* Participation in brain stimulation within the past 3 months
* Regular use of walking aid
* Significant Tai Chi experience (> 6 months training in past 2 years)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Rate of participant recruitment | 24 months
Protocol adherence | 6 months
  The percentage of Tai Chi classes attended and home practice completed by each participant randomized to the experimental arm.
Retention | 6 months
  The percentage of study visits completed by each participant.

SECONDARY OUTCOMES:
Change from Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline and 6 months
  Motor symptom severity
Change from Baseline in PDQ-39 | Baseline and 6 months
  PD-related quality of life
Change from Baseline in Physical Activity Status Scale (PASS) | Baseline and 6 months
Change from Baseline in Self-Efficacy for Exercise Scale | Baseline and 6 months
Change from Baseline in Activity-specific Balance Confidence Scale | Baseline and 6 months
Change from Baseline in Profile of Mood State | Baseline and 6 months
Change from Baseline in Single leg stance time | Baseline and 6 months
Change from Baseline in Timed Up and Go Test | Baseline and 6 months
Change from Baseline in Steady state gait dynamics | Baseline and 6 months
  Steady state gait dynamics during 90 seconds of continuous over ground walking at preferred speed with and without use of dual task challenges
Change from Baseline in Balance/Postural control | Baseline and 6 months
  Sway based measures of balance during quiet and tandem standing, with and without dual tasks
Change from Baseline in Cognitive function | Baseline and 6 months
  Trail Making Test (TMT), The Digit Span Test, Controlled Oral Word Association Test (COWAT), Stroop Color-Word Test

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Wayne, PhD, Principal Investigator — Harvard University Faculty of Medicine
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886